CLINICAL TRIAL: NCT04643262
Title: Sleeve Gastrectomy: Outcome, Morbidity and Mortality. A Multicentric Retrospective Trial. PSICHE TRIAL (Postoperative Sleevegastrectomy Italian or (International) Group Complications Highlights Experience)
Brief Title: Sleeve Gastrectomy: Outcome, Morbidity and Mortality. A Multicentric Retrospective Trial
Acronym: PSICHE
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, MD,PhD, Responsible for the Bariatric and Metabolic Surgery unit, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 18112010
Record Dates: First submitted 2020-11-13; First posted 2020-11-25 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Morbid Obesity
Keywords: Bariatric surgery; morbidity and mortality
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intraoperative morbidity and mortality: Intraoperative complications (i.e. splenectomy, bleeding, positive leak test if performed) and type treatment are collected and recorded.
  Interventions: Procedure: Sleeve Gastrectomy
- peri-operative morbidity and mortality (<30 days): Perioperative complications (<30 days) considered are mortality, morbidity (i.e. leak, bleeding, occlusion, pneumonia, vascular complications, portal pulmonary-splenic embolism) and type treatment.
  Interventions: Procedure: Sleeve Gastrectomy
- Post-operative morbidity and mortality (>30 days): Postoperative complications (>30 days) considered are morbidity, mortality (i.e. leak, embolism, Incisional trocar hernia, other) and type treatment
  Interventions: Procedure: Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Sleeve Gastrectomy — Once the left crus is reached, an optimal exposure of the hiatus is mandatory to find incidental hiatal hernias and a complete dissection of the left crus performed to prevent retained fundus. The greater omentum was opened close to the stomach wall in some part in between the fundus and the antrum to have greater curvature completely detached from the stomach; this dissection starts at 2 cm or _____proximal to the pylorus and continued along the greater curvature to the left crus. Posterior adhesions if present, were carefully divided. The left gastrophrenic ligament was divided to expose the angle of His to identify the complete hiatus and fundus. A bougie was positioned before starting resection of the stomach. We use a 36French bougie or --------- we have chosen cartridges Black at the antrum level and finished with a purple cartridge. We always checked the posterior wall before firing.

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) is currently the most frequent primary bariatric procedure performed worldwide. LSG is a safe and effective technique in terms of excess weight loss and it is, moreover, a powerful metabolic operation that activates significant hormonal pathways that lead to changes in eating behavior, glycemic control and intestinal functions.Regarding a technical point of view, LSG might be considered a time saving procedure for the absence of intestinal anastomosis. The most frequent and sometimes dangerous complications are leaking, hemorrhage, splenic injury, stenosis and Gastro-Esophageal Reflux Disease (GERD). Despite its established efficacy and safety, dispute still exists on the optimal conduction of LSG operative technique: bougie size, distance of resection margin from the pylorus, the shape of section at the gastroesophageal junction, staple line reinforcement and intraoperative leak testing are among the most controversial issues .

Thus, the primary aim of the present retrospective multicentric study is to evaluate intra and peri-operatory (< 30 days) and post-operative (> 30 days) morbidity and mortality rates of patients undergone LSG, and the correlation of the latter rates with different surgical measures. Secondary aim is to evaluate the strategy for the treatment of the complication, and if there is a correlation between morbidity/mortality and volume of the Bariatric Center

DETAILED DESCRIPTION:
This study is a retrospective multicenter trial conduct from January 2015 to December 2020 in 10 centers. All the procedures were performed by the (---- number of surgeons). Morbid obesity was preoperatively diagnosed according to the International Federation for Surgery of Obesity (IFSO) guidelines. Patients were collected in a electronic database and categorized according to the following parameters:

* Distance of resection margin from the pylorus (>5 cm / <5 cm)
* Bougie size (>34 French, <34 French)
* Distance of resection margin from the gastroesophageal junction (>…cm/<...cm)
* Staple line reinforcement (Yes/No - If yes, the reinforcement technique will be reported)
* Intraoperative leak testing (Yes/No - If yes, the test used will be reported)
* Number and size of trocar used and access closure technique (Yes/No - If yes, the technique will be reported) The study protocol was approved by the regional Ethics Committee. 2.2 Inclusion criteria Inclusion criteria were morbid obesity defined as BMI 40 kg/m2 or BMI>35 with comorbidity and age between 25-60 years old. Obesity-related comorbidities included Type 2 Mellitus Diabetes (T2MD), hypertension, hyperlipidemia, bronchial asthma, osteoarthritis and degenerative joint disease.

2.3 Exclusion Criteria Patients with endocrine disorders causing obesity (as hypothyroidism and Cushing disease), pregnancy or lactation, psychiatric illness, or recent diagnosis of malignancy, inflammatory bowel disease, Barrett ́s esophagus, and GERD with esophagitis scored as or greater than grade B, a large hiatal hernia (>3 cm) were excluded from the study.

2.4 Study Outcomes The primary aims of the present retrospective multicentric study is to evaluate intra and peri and post operatory morbidity and mortality rates (< 30 and >30 days) of patients undergone Laparoscopic Sleeve Gastrectomy, and the correlation of the latter rates with different surgical measures. Secondary aims is to evaluate the strategy for the treatment of the complication, and if there is a correlation between morbidity/mortality and the volume of the Bariatric Center.

2.6 Blinding Process Physicians and staff who will collect the data and those who will evaluate the endpoints will all be unaware of the patients allocation. Patients will be collected in an electronic database with consecutive numbers without the possibility of identifying the center of origin until the final evaluation of the study endpoints. As the blinding process for the operating surgeons is not feasible, they are not involved in data collection and evaluation of results.

2.5 Pre-operative evaluation Preoperative evaluation included anthropometric measurements (height in cm, weight in kg, Body Mass Index (BMI) in kg/m2), comorbidity evaluation [Glycated Hemoglobin(A1c), C-peptide, stimulated C-peptide, Electrocardiography (ECG), echocardiography, lower limbs US color-doppler study, thyroid function profile]. All patients were evaluated for the presence/absence of Gastro Esophageal Reflux Disease before surgery through a preoperative upper endoscopy with an eventual esophageal biopsy. The presence of helicobacter pylori is also investigated with for a rapid urease test on an antral specimen.

2.7 Surgical Technique The patient is placed in a split leg position with the surgeon located in between the patient's legs. Closed pneumoperitoneum was established using our standard technique of Verres needle insufflation in Palmer site and optical insertion of a 12-mm port at a supraumbilical site (10-15 cm from umbilicus) Two further 15-mm and 12-mm ports were placed respectively in the left and right ipocondrum as working ports. A subxiphoid track was created using a 5-mm port for placement of a liver retractor. In patients with higher body mass index who have severe visceral obesity, additional trocars can be added for retraction of the omentum or big fatty livers, to optimize the exposure to reach the left crus. Once the left crus is reached, an optimal exposure of the hiatus is mandatory to find incidental hiatal hernias and a complete dissection of the left crus performed to prevent retained fundus. The greater omentum was opened close to the stomach wall in some part in between the fundus and the antrum to have greater curvature completely detached from the stomach; this dissection starts at 2 cm or _____proximal to the pylorus and continued along the greater curvature to the left crus. Posterior adhesions if present, were carefully divided. The left gastrophrenic ligament was divided to expose the angle of His to identify the complete hiatus and fundus. A bougie was positioned before starting resection of the stomach. Researchers use a 36French bougie or --------- Researchers have chosen cartridges Black at the antrum level and finished with a purple cartridge. Researchers always checked the posterior wall before firing. Once Researchers have reached the proximal stomach, the stapler has to be positioned 1 cm lateral to the left of the angle of His to avoid inclusion of esophageal tissue. Methylene blue test is performed routinely.

2.8 Post-operative evaluation Regarding the primary endpoints, intraoperative complications (i.e. splenectomy, bleeding, positive leak test if performed) and type treatment are collected and recorded. Perioperative complications (<30 days) considered are mortality, morbidity (i.e. leak, bleeding, occlusion, pneumonia, vascular complications, portal pulmonary-splenic embolism) and type treatment. Postoperative complications (>30 days) considered are morbidity, mortality (i.e. leak, embolism, Incisional trocar hernia, other) and type treatment Regarding the secondary endpoint, in case of gastric fistula onset its diagnosis method (clinical, instrumental) and its management (timing, surgical or endoscopic - endoprosthesis, pigtails, clips-) or both) are collected and recorded. In case of postoperative bleeding, its diagnosis method (clinical, instrumental) and its management (timing, Surgical, medical) are collected and recorded.

3.6 Statistical Analysis Continuous data are expressed as median and interquartile (25-75th) range or mean and Standard Deviation (SD), unless otherwise indicated. Differences between preoperative and postoperative parameters were compared by Wilcoxon paired rank test. Median time of follow-up was estimated using the Kaplan-Meier method. Multivariable analysis was conducted through a forward-backward stepwise Cox regression based on Akaike Information Criterion (AIC) considering age, gender, % Excess Weighth Loss, Body Mass Index and treatment.

For all tests, the cut-off for statistical significance was set at p= 0.05. Statistical analysis was performed using R v3.5.0.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity defined as Body Mass Index 40 kg/m2
* Body Mass Index >35 with comorbidity (Type 2 Mellitus Diabetes (T2MD), hypertension, hyperlipidemia, bronchial asthma, osteoarthritis))
* Age between 25-68 years old.

Exclusion Criteria:

* Patients with endocrine disorders causing obesity (as hypothyroidism and Cushing disease)
* Pregnancy or lactation
* Psychiatric illness
* Recent diagnosis of malignancy
* Inflammatory bowel disease
* Barrett ́s esophagus

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective multicenter trial conduct from January 2015 to December 2020 in 20 centers. All patients underwent Sleeve Gastrectomy. All the procedures were performed by the (---- number of surgeons). Morbid obesity was preoperatively diagnosed according to the International Federation for Surgery of Obesity (IFSO) guidelines
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative complications | time 0
  splenectomy, bleeding, positive leak test if performed
Perioperative complications | up to 4 weeks from surgery
  Mortality
Perioperative complications | up to 4 weeks from surgery
  Morbidity:( leak, bleeding, occlusion, pneumonia, vascular complications, portal pulmonary-splenic embolism) < 30 days
Postoperative complications | up to 6 months
  Mortality
Postoperative complications | up to 6 months
  Morbidity: (leak, embolism, Incisional trocar hernia) >30 days